CLINICAL TRIAL: NCT06940011
Title: Glycocalyx Restoration in Treatment Resistant Hypertension: a Proof of Concept, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Endocalyx in Treatment Resistent Hypertension
Acronym: GLYCO-TRH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Heart Foundation (Other); Dutch Kidney Foundation (Other); Microvascular Health Solutions LLC (Unknown)
Responsible Party: Principal Investigator, Rik Olde Engberink, Principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL85685.018.24
Record Dates: First submitted 2025-01-20; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Treatment Resistant Hypertension
Keywords: Glycocalyx; Glycosaminoglycans; non-osmotic sodium storage; hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endocalyx Pro (Experimental): Endocalyx is a food supplement that is distributed by Microvascular Health Solutions LLC in Chattanooga, Tennessee. Patients will receive 4 capsules Endocalyx per day, for 12 consecutive weeks. The capsules are orally administered and can be taken with water, on an empty stomach or with food. If possible, the patient will take 2 capsules in the morning, and 2 capsules in the afternoon. If preferred by the patient, the 4 capsules could also be taken once daily in the morning.
  Interventions: Dietary Supplement: Endocalyx Pro
- Placebo (Placebo Comparator): Placebo pills will be provided by Microvascular Health Solutions and are matched with the Endocalyx capsules. The placebo capsules contain no active pharmaceutical ingredients and contain solely widely used excipients. Patients will receive 4 capsules of the placebo per day for 12 consecutive weeks. The capsules are orally administered and can be taken with water, on an empty stomach or with food. If possible, the patient will take 2 capsules in the morning, and 2 capsules in the afternoon. If preferred by the patient, the 4 capsules could also be taken once daily in the morning.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Endocalyx Pro — 4 capsules once daily OR 2 capsules twice daily
  Arms: Endocalyx Pro
Other: Placebo — 4 capsules once daily OR 2 capsules twice daily
  Arms: Placebo

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled study is to assess whether the food supplement Endocalyx lowers blood pressure in patients with treatment resistant hypertension.

DETAILED DESCRIPTION:
During this intervention study, subjects will receive either a placebo or Endocalyx for 12 weeks. The main objective of this study is to assess whether the food supplement Endocalyx lowers blood pressure in patients with treatment resistant hypertension.

Secondary objectives are:

* Change from baseline in office blood pressure and 24-hour blood pressure profiles in subjects with treatment resistant hypertension.
* To assess whether sodium intake, sex or kidney function modulates the effect of Endocalyx on blood pressure.
* Change from baseline in total vessel density, perfused vessel density, proportion of perfused vessels and microvascular health score
* To assess the effect of Endocalyx on total peripheral resistance.
* The effect of Endocalyx on quality of life.
* To estimate the potential impact of Endocalyx on long-term cardiovascular protection and health care costs.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment resistant hypertension defined as

   1. an uncontrolled office BP (≥140/90 mmHg).
   2. is on a regimen of ≥3 adequately dosed antihypertensive agents of different classes, including a diuretic, at maximum tolerated dose based on investigator judgment.
2. Stable diuretic and antihypertensive treatment for the previous 3 weeks.
3. Subject, or legal representative, has voluntarily signed and dated an Informed Consent Form, approved by the Independent Ethics Committee (IEC).

Exclusion Criteria:

1. Age <18 years.
2. Estimated glomerular filtration rate (eGFR) <20 ml/min/1.73m2 measured by the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine formula and the 2012 cystatin C CKD-EPI formula.
3. A mean seated systolic blood pressure of at least 180 mmHg or a diastolic blood pressure of at least 110 mmHg.
4. Known secondary hypertension
5. An acute coronary syndrome, stroke, transient ischemic attack or cardiovascular surgery in the last 3 months.
6. Hospitalization for heart failure in the past 3 weeks.
7. Dialysis treatment or expected initiation of dialysis within 3 months of screening.
8. Women of child bearing potential who are not taking adequate contraception (i.e. <1% failure rate).
9. Planned surgery in the next 12 weeks
10. Major surgery in the previous 4 weeks.
11. Use of prednisolone >5 mg/day
12. Use of any other investigational drug.
13. Presence of significant comorbidities (e.g., advanced malignancy, advanced liver disease) with a life expectancy of less than 1 year.
14. A psychiatric, addictive or any disorder that compromises ability to give truly informed consent for participation in this study.
15. Known hypersensitivity to seaweed, corn, artichoke, grape, melon or to any of the excipients of Endocalyx.
16. Known hypersensitivity or allergies for milk, eggs, fish, crustacean shellfish, tree nuts, peanuts, wheat and soybeans.
17. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose galactose malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 24-hour systolic blood pressure | 12 weeks
  We will perform an uncorrected analysis and an analysis that is corrected for the reported and measured changes in antihypertensive medication use.

SECONDARY OUTCOMES:
Change from baseline in 24-hour diastolic blood pressure | 12 weeks
Change from baseline in seated systolic office blood pressure | 12 weeks
Change from baseline in seated diastolic office blood pressure | 12 weeks
Change from baseline in percentage of patients with a night-time blood pressure dip | 12 weeks
  The nighttime blood pressure dipping status will be measured with a 24-hour blood pressure measurements. Patients will be classified as a 'dippers' when the nighttime systolic blood pressure and/or diastolic blood pressure falls >10% and <20% compared to daytime readings. Exteme dippers are described as those with blood pressure fall of at least 20%. Patients with blood pressure fall between 0 and 10% are classified as non-dippers.
Percentage of patients achieving a seated office blood pressure <140/90 mmHg after intervention | 12 weeks
  Participants achieved a response if the systolic blood pressure is below 140 mmHg and the diastolic blood pressure is below 90 mmHg
Percentage of patients that needed additional antihypertensive drugs and/or higher dosage of antihypertensive drugs during the study | 12 weeks
Percentage of patients that required lowering of their antihypertensive drugs during the study | 12 weeks
Change from baseline in total vessel density and perfused vessel density | 12 weeks
  The total vessel density and perfused vessel density will be measured using Sidestream Dark Field imaging.
Change from baseline in proportion of perfused vessels | 12 weeks
  The proportion of perfussed vessels will be measured using Sidestream Dark Field imaging.
Change from baseline in microvascular flow index | 12 weeks
  The microvascular flow index will be measured using Sidestream Dark Field imaging.
Change from baseline in microvascular health score | 12 weeks
  The microvascular health score will be measured using Sidestream Dark Field imaging.
Change from baseline in heart rate | 12 weeks
  The heart rate will be measured using the Nexfin device
Change from baseline in total peripheral resistance | 12 weeks
  The total pheripheral resistance will be measured using the Nexfin device
Change from baseline in cardiac output | 12 weeks
  The cardiac output will be measured using the Nexfin device
Change from baseline in quality of life | 12 weeks
  Quality of life will be evaluated by the SF-36 questionnaire.
The potential impact of Endocalyx on long-term cardiovascular protection and health care costs. | 12 weeks
  The EQ-5D-5L questionnaire will be used to score a patient health status and will be transposed in quality adjusted life years (QALY's).
Change from baseline in skin sodium content | 12 weeks
  Skin sodium content will measured using a 7T sodium MRI
Change from baseline in muscle sodium content | 12 weeks
  Muscle sodium content will measured using a 7T sodium MRI
Change from baseline in skin water content | 12 weeks
  Skin water content will measured using a 7T H-MRI
Change from baseline in muscle water content | 12 weeks
  Muscle water content will measured using a 7T H-MRI
Change from baseline in transepidermal water loss | 12 weeks
  Transepidermal water loss will be measured with the Tewameter® TM Hex probe
Change from baseline in skin hydration | 12 weeks
  The skin hydration will be measured using the Corneometer® CM 825 probe
Change from baseline in total body water | 12 weeks
  The change in total body water (liter) will be measured using the bioelectrical impendance analysis
Incidence of adverse events in the Endocalyx group compared to the placebo group | 12 weeks

OTHER OUTCOMES:
To assess whether sodium intake, measured using 24-hour urine collection, modulate the effect of Endocalyx on blood pressure. | 12 weeks
  We will study the (possible) modulatory effect sodium intake (mmol/L), measuring using 24 hours urine collection, on the effect of endocalyx on blood pressure.
To assess whether sex modulate the effect of Endocalyx on blood pressure. | 12 weeks
  The association between sex and the effect of endocalyx on blood pressure.
To assess whether kidney function modulate the effect of Endocalyx on blood pressure. | 12 weeks
  The association between kidney function and the effect of endocalyx on blood pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researcher